CLINICAL TRIAL: NCT02374840
Title: Pharmacogenomics Registry to Assess Clinical Utility
Acronym: PREACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Companion Dx Reference Lab, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CD-2014-102
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Drug Side Effects
Keywords: Pharmacogenomics; Adverse Drug Reactions; Pharmacogenetics
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The PREACT Registry aims to see whether data from Pharmacogenomic Testing (PGx) can help healthcare providers manage patient medication regimens and assess if the testing has an effect on reducing medication side effects, hospitalizations and emergency department visits.

The way an individual processes a drug is in part determined by their genes, and there is known to be genetic variation between humans in the way drugs are metabolized. The study of the way genes affect a person's response to drugs is known as "Pharmacogenomics."

ELIGIBILITY:
Inclusion Criteria:

* Pharmacogenomic testing has been performed within 12-months prior to eligibility assessment for genes known to influence metabolism of at least one target drug
* Subject is 2 years of age or older
* Subject is not taking an investigational medication or in a clinical trial that would interfere with participation in the registry

Exclusion Criteria:

* Subject's medical and medication history is unavailable over the 90-day period preceding the receipt of pharmacogenomic test results
* Subject (or subject's parent/guardian) is unable to provide an accurate history due to mental incapacity, in the Investigator's opinion.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects aged 2 years and above, currently receiving or under consideration to receive at least one medication known to be metabolized through relevant genetically-modified pathways.
Sampling Method: Non-Probability Sample
Enrollment: 340778 (Estimated)
Dates: Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Meaningful Change | 90 day
  Binary occurrence of meaningful change in drug regimen, defined for each subject as:
  * A genotype known to affect a target drug is identified by pharmacogenomic testing, and
  * The treating physician makes at least one target drug regimen change in dose, frequency, route of administration, drug discontinuation, addition or substitution.

SECONDARY OUTCOMES:
Changes in target drug regimen | 90 days retrospective; 90 days prospective
  Changes in target drug regimen over the 90-day period preceding receipt of PGx results, compared to the changes made in the 90-day period thereafter.
Number of target drug adverse events (TDAE) | 90 day retrospective; 90 day prospective
  Number of TDAE over the 90-day period preceding receipt of pharmacogenomics test results compared with the number over the 90-day period after the test
Target drug related emergency department visits | 90 day retrospective; 90 day prospective
  Emergency department visits over the 90-day period prior to receipt of pharmacogenomics test results, compared to the number of visits over the 90-day period following receipt of test results.
Target drug related hospitalizations | 90 day retrospective; 90 day prospective
  Hospitalizations over the 90-day period prior to receipt of pharmacogenomics test results, compared to the number of visits over the 90-day period following receipt of test results.